CLINICAL TRIAL: NCT00297661
Title: Sirolimus-Eluting Versus Paclitaxel-Eluting Stents for Coronary Revascularization: SIRTAX Trial
Brief Title: Sirolimus-Eluting Versus Paclitaxel-Eluting Stents for Coronary Revascularization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KEK-33/2003
Record Dates: First submitted 2006-02-22; First posted 2006-02-28 (Estimated); Last update posted 2006-10-20 (Estimated); Status verified 2006-02

CONDITIONS: Coronary Heart Disease
Keywords: Coronary Revascularization; Sirolimus-eluting stents; Paclitaxel-eluting stents
MeSH Terms: conditions — Coronary Disease

INTERVENTIONS:
Device: Sirolimus-eluting stent
Device: Paclitaxel-eluting stent

SUMMARY:
Context: Sirolimus-eluting stents and paclitaxel-eluting stents, as compared with bare-metal stents, reduce the risk of restenosis. It is unclear whether there are differences in safety and efficacy between the two types of drug-eluting stents.

Objective: To determine differences in safety and efficacy between sirolimus and paclitaxel eluting stents.

DETAILED DESCRIPTION:
Design: Randomized controlled, observer-blind trial comparing sirolimus-eluting stents with paclitaxel-eluting stents

Patients: 1012 patients undergoing percutaneous coronary intervention. The two groups had similar baseline clinical and angiographic characteristics.

ELIGIBILITY:
Inclusion Criteria:

Patients with either stable angina or an acute coronary syndrome were eligible to participate if they had at least one lesion with stenosis of at least 50 percent in a vessel with a reference diameter between 2.25 and 4.00 mm that was suitable for stent implantation.

Exclusion Criteria:

Allergy to antiplatelet drugs, heparin, stainless steel, contrast agents, sirolimus, or paclitaxel; participation in another coronary-device study; and terminal illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1012
Dates: Start 2003-04

PRIMARY OUTCOMES:
Major adverse cardiac events at nine months (composite of cardiac death, myocardial infarction or ischemia-driven target lesion revascularization)

SECONDARY OUTCOMES:
Clinical: Ischemia-driven target lesion revascularization, target-vessel revascularization, and target-vessel failure (composite of cardiac death, myocardial infarction or ischemia-driven target-vessel revascularization)
Angiographic: In-segment late luminal loss

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Windecker, MD, Principal Investigator — Department of Cardiology, University Hospital Bern; Peter Juni, MD, Study Director — Department of Social and Preventive Medicine, University of Bern; Bernhard Meier, MD, Study Chair — Department of Cardiology, University Hospital Bern
Locations (1):
- University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Result] Windecker S, Remondino A, Eberli FR, Juni P, Raber L, Wenaweser P, Togni M, Billinger M, Tuller D, Seiler C, Roffi M, Corti R, Sutsch G, Maier W, Luscher T, Hess OM, Egger M, Meier B. Sirolimus-eluting and paclitaxel-eluting stents for coronary revascularization. N Engl J Med. 2005 Aug 18;353(7):653-62. doi: 10.1056/NEJMoa051175. Epub 2005 Aug 16. PMID 16105989
- [Derived] Yamaji K, Raber L, Zanchin T, Spitzer E, Zanchin C, Pilgrim T, Stortecky S, Moschovitis A, Billinger M, Schonenberger C, Eberli F, Juni P, Luscher TF, Heg D, Windecker S. Ten-year clinical outcomes of first-generation drug-eluting stents: the Sirolimus-Eluting vs. Paclitaxel-Eluting Stents for Coronary Revascularization (SIRTAX) VERY LATE trial. Eur Heart J. 2016 Dec 1;37(45):3386-3395. doi: 10.1093/eurheartj/ehw343. Epub 2016 Aug 30. PMID 27578808
- [Derived] Koskinas KC, Siontis GC, Piccolo R, Franzone A, Haynes A, Rat-Wirtzler J, Silber S, Serruys PW, Pilgrim T, Raber L, Heg D, Juni P, Windecker S. Impact of Diabetic Status on Outcomes After Revascularization With Drug-Eluting Stents in Relation to Coronary Artery Disease Complexity: Patient-Level Pooled Analysis of 6081 Patients. Circ Cardiovasc Interv. 2016 Feb;9(2):e003255. doi: 10.1161/CIRCINTERVENTIONS.115.003255. PMID 26823484
- [Derived] Vranckx P, Kalesan B, Stefanini GG, Farooq V, Onuma Y, Silber S, de Vries T, Juni P, Serruys PW, Windecker S. Clinical outcome of patients with stable ischaemic heart disease as compared to those with acute coronary syndromes after percutaneous coronary intervention. EuroIntervention. 2015 Jun;11(2):171-9. doi: 10.4244/EIJV11I2A31. PMID 24531331
- [Derived] Stefanini GG, Kalesan B, Pilgrim T, Raber L, Onuma Y, Silber S, Serruys PW, Meier B, Juni P, Windecker S. Impact of sex on clinical and angiographic outcomes among patients undergoing revascularization with drug-eluting stents. JACC Cardiovasc Interv. 2012 Mar;5(3):301-10. doi: 10.1016/j.jcin.2011.11.011. PMID 22440496
- [Derived] Girasis C, Garg S, Raber L, Sarno G, Morel MA, Garcia-Garcia HM, Luscher TF, Serruys PW, Windecker S. SYNTAX score and Clinical SYNTAX score as predictors of very long-term clinical outcomes in patients undergoing percutaneous coronary interventions: a substudy of SIRolimus-eluting stent compared with pacliTAXel-eluting stent for coronary revascularization (SIRTAX) trial. Eur Heart J. 2011 Dec;32(24):3115-27. doi: 10.1093/eurheartj/ehr369. Epub 2011 Sep 27. PMID 21951630
- [Derived] Raber L, Wohlwend L, Wigger M, Togni M, Wandel S, Wenaweser P, Cook S, Moschovitis A, Vogel R, Kalesan B, Seiler C, Eberli F, Luscher TF, Meier B, Juni P, Windecker S. Five-year clinical and angiographic outcomes of a randomized comparison of sirolimus-eluting and paclitaxel-eluting stents: results of the Sirolimus-Eluting Versus Paclitaxel-Eluting Stents for Coronary Revascularization LATE trial. Circulation. 2011 Jun 21;123(24):2819-28, 6 p following 2828. doi: 10.1161/CIRCULATIONAHA.110.004762. Epub 2011 Jun 6. PMID 21646500
- [Derived] Raber L, Juni P, Loffel L, Wandel S, Cook S, Wenaweser P, Togni M, Vogel R, Seiler C, Eberli F, Luscher T, Meier B, Windecker S. Impact of stent overlap on angiographic and long-term clinical outcome in patients undergoing drug-eluting stent implantation. J Am Coll Cardiol. 2010 Mar 23;55(12):1178-1188. doi: 10.1016/j.jacc.2009.11.052. PMID 20298923
- [Derived] Billinger M, Beutler J, Taghetchian KR, Remondino A, Wenaweser P, Cook S, Togni M, Seiler C, Stettler C, Eberli FR, Luscher TF, Wandel S, Juni P, Meier B, Windecker S. Two-year clinical outcome after implantation of sirolimus-eluting and paclitaxel-eluting stents in diabetic patients. Eur Heart J. 2008 Mar;29(6):718-25. doi: 10.1093/eurheartj/ehn021. Epub 2008 Feb 12. PMID 18272504
- [Derived] Togni M, Eber S, Widmer J, Billinger M, Wenaweser P, Cook S, Vogel R, Seiler C, Eberli FR, Maier W, Corti R, Roffi M, Luscher TF, Garachemani A, Hess OM, Wandel S, Meier B, Juni P, Windecker S. Impact of vessel size on outcome after implantation of sirolimus-eluting and paclitaxel-eluting stents: a subgroup analysis of the SIRTAX trial. J Am Coll Cardiol. 2007 Sep 18;50(12):1123-31. doi: 10.1016/j.jacc.2007.06.015. Epub 2007 Sep 4. PMID 17868802